CLINICAL TRIAL: NCT04377984
Title: Impact of a Strategy Combining Morphine Savings and a Loco-regional Anesthesia Technique on the Quality of Post-operative Rehabilitation of Cesareans Performed Under Peri-spinal Anesthesia
Brief Title: Impact of a Strategy Combining Morphine Savings and Anesthesia Technique on the Quality of Post-operative Rehabilitation
Acronym: REHACESAR
Status: Terminated | Type: Observational
Why Stopped: Because of health context as well as the implementation of the RAAC caesarean section, which means that patients enter in the morning, and it is therefore no longer possible to do the QOR on D-1 and therefore to include scheduled caesarean sections
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-09Obs-CHRMT
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-09

CONDITIONS: Cesarean Section Complications
Keywords: cesarean; anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of REHACESAR is to study the impact of an association of a low dose of neuraxial morphine and a locoregional anesthesia (TAP block or catheter for continuous wound infiltration) on quality of recovery after cesarean delivery under regional anesthesia.

To assess the quality of recovery, women complete the self-questionnaire Quality Of Recovery (QOR)15 on D-1 (the day before cesarean, if elective), D+1, +2 and +3 after surgery.

The QOR-15 is a 15 items questionnaire which provides a valid and efficient evaluation of the postoperative quality of recovery.

REHACESAR is a prospective observational study. It takes place in the maternity of the CHR Metz-Thionville hospital.

DETAILED DESCRIPTION:
Cesarean delivery is a very frequent surgical procedure. In France 20,4% of all births occur by cesarean section. Regional anesthesia (Spinal or epidural anesthesia) is the most common type of anesthesia for emergent or elective cesarean section.

HAS guidelines on Enhanced Recovery After Surgery (ERAS) include cesarean section. ERAS is a "multimodal perioperative care pathway designed to achieve early recovery for patients undergoing surgery". The aim is to avoid factors which delay recovery: nausea and vomiting, pain, postoperative ileus…

Postoperative analgesia is a key factor in ERAS because pain may prolong recovery and has a negative impact on rehabilitation. Among the multimodal analgesia we can use neuraxial morphine: epidural or intrathecal. Neuraxial morphine is effective for post-cesarean analgesia. Previous studies have attempted to determine the optimum intrathecal and epidural morphine doses. The aim is to provide the better analgesia with fewer side effects (pruritus, nausea and vomiting, ileus) Another way to provide analgesia is locoregional anesthesia: continuous wound infiltration and Transversus Abdominis Plane Block (TAP) block.

The aim of REHACESAR is to study the impact of an association of a low dose of neuraxial morphine and a locoregional anesthesia (TAP block or catheter for continuous wound infiltration) on quality of recovery after cesarean delivery under regional anesthesia.

To assess the quality of recovery, women complete the self-questionnaire Quality Of Recovery (QOR)15 on D-1 (the day before cesarean, if elective), D+1, +2 and +3 after surgery.

The QOR-15 is a 15 items questionnaire which provides a valid and efficient evaluation of the postoperative quality of recovery.

REHACESAR is a prospective observational study. It takes place in the maternity of the CHR Metz-Thionville hospital.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman,
* operated on a scheduled cesarean under spinal anesthesia or urgent under epidural anesthesia, with use of perimedullary morphine

Exclusion Criteria:

* Contraindication to the use of morphine
* Contraindication to local anesthetics
* Urgent cesarean section for maternal pathology: preeclampsia (PE), eclampsia, HELLP syndrome
* Post-operative maternal transfer
* Preoperative opiate treatment
* Patient unable to understand and / or answer a questionnaire in French

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant woman operated on a scheduled cesarean under spinal anesthesia or urgent under epidural anesthesia, with use of perimedullary morphine
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the QOR-15 D1 post-caesarean score between six different groups | day1
  The QoR 15 score is a score of 15 items, each scored from 0 to 10. These items assess 5 dimensions of post-operative recovery: pain, physical comfort, functional autonomy, emotions and psychological support.
  These 15 items represent the quality of post-operative rehabilitation in its physical and mental dimensions

SECONDARY OUTCOMES:
Comparison between the different anesthesia groups of the post-operative period before resumption of gastrointestinal transit. | day 3
  The corresponding criterion will be the time in hours between surgery and the resumption of a gas transit

CONTACTS AND LOCATIONS:
Overall Officials: Julien Nadaud, Principal Investigator — CHR Metz Thionville
Locations (1):
- CHR Metz-Thionville, Metz, France